CLINICAL TRIAL: NCT03045328
Title: An Open Label Phase 2 Trial of Venetoclax With Ibrutinib in Relapsed or Refractory Chronic Lymphocytic Leukemia and Small Lymphocytic Lymphoma
Brief Title: Venetoclax and Ibrutinib in Patients With Relapsed/Refractory CLL or SLL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Steven E. Coutre (Other)
Responsible Party: Sponsor-Investigator, Steven E. Coutre, Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-36705; NCI-2017-00124 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HEM0048 (Other: OnCore)
Record Dates: First submitted 2017-02-03; First posted 2017-02-07 (Estimated); Results first posted 2021-09-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Recurrent Chronic Lymphocytic Leukemia; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ibrutinib, venetoclax) (Experimental): Patients receive ibrutinib PO QD beginning on week 1 day 1. Treatment with ibrutinib continues in the absence of disease progression or unacceptable toxicity. Patients also receive venetoclax PO QD beginning on week 9 day 1. Treatment with venetoclax continues up to week 61 day 7 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Drug: Venetoclax

INTERVENTIONS:
Drug: Ibrutinib — Administered at 420 mg/day, as oral capsules (3 x 140 mg), starting Day 1, Week 1.
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Drug: Venetoclax — Administered as tablets, starting Day 1, Week 9, with dose increasing every 7 days through 5 dose levels (20 mg; 50 mg; 100 mg; 200 mg; 400 mg).
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta

SUMMARY:
This is an open-label non-randomized two-center phase 2 study evaluating the safety and efficacy of concurrent therapy with ibrutinib and venetoclax in subjects with relapsed or refractory CLL/SLL.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy of concurrent therapy with ibrutinib and venetoclax in patients with relapsed and refractory chronic lymphocytic leukemia (CLL) and small lymphocytic leukemia (SLL).

The secondary objectives of this study are to define the safety, tolerability, and dose-limiting toxicity (DLT) within 28 days of completion of dose-escalation.

ELIGIBILITY:
Inclusion Criteria:

* Subject must voluntarily sign and date an informed consent approved by the Institutional Review Board prior to initiation of any study specific procedures
* Subject must have a diagnosis of CLL that meets International Workshop on Chronic Lymphocytic Leukemia (IWCLL)/National Cancer Institute (NCI)-Working Group (WG) criteria
* Subject must have relapsed/refractory disease with an indication for treatment according to the 2008 IWCLL/NCI WG criteria
* Measurable nodal disease by computed tomography (CT)
* Absolute neutrophil count > 750 cells/mm^3 (0.75 x 10^9/L)
* Platelet count > 30,000 cells/mm^3 (30 x 10^9/L)
* Hemoglobin > 8.0 g/dL
* Serum aspartate transaminase (AST) or alanine transaminase (ALT) =< 2.5 x upper limit of normal (ULN)
* Estimated creatinine clearance >= 30 mL/min (Cockcroft-Gault)
* Bilirubin =< 1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin)
* Prothrombin time/international normalized ratio (PT/INR) < 1.5 x ULN and partial thromboplastin time (PTT) (activated [a]PTT) < 1.5 x ULN
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Female subjects who are of non-reproductive potential (ie, post-menopausal by history - no menses for >= 1 year; OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy); female subjects of childbearing potential must have a negative serum pregnancy test upon study entry
* Male and female subjects must agree to use highly effective methods of birth control (eg, condoms, implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], sexual abstinence, or sterilized partner) during the period of therapy and for 90 days after the last dose of study drug

Exclusion Criteria:

* Subject has previously received either venetoclax or ibrutinib
* Subject has received a live virus vaccine within 28 days prior to the initiation of study treatment
* Subject has undergone an allogeneic stem cell transplant in the past 1 year and must not have active chronic graft versus host disease (cGVHD) if over 1 year post allogeneic transplant
* Subject has developed Richter's transformation confirmed by biopsy
* Chemotherapy =< 21 days prior to first administration of study treatment and/or monoclonal antibody =< 6 weeks prior to first administration of study treatment
* History of other malignancies, except:

  * Malignancy treated with curative intent and with no known active disease present for >= 3 years before the first dose of study drug and felt to be at low risk for recurrence by treating physician
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
* Concurrent systemic immunosuppressant therapy (eg, cyclosporine A, tacrolimus, etc, or chronic administration [> 14 days] of > 20 mg/day of prednisone) within 28 days of the first dose of study drug
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug
* Recent infection requiring systemic treatment that was completed =< 14 days before the first dose of study drug
* Unresolved toxicities from prior anti-cancer therapy, defined as having not resolved to Common Terminology Criteria for Adverse Event (CTCAE, version [v]4), grade =< 1, or to the levels dictated in the inclusion/exclusion criteria with the exception of alopecia
* Known bleeding disorders (eg, von Willebrand's disease) or hemophilia
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment
* Known history of human immunodeficiency virus (HIV) or active with hepatitis C virus (HCV) or hepatitis B virus (HBV); subjects who are positive for hepatitis B core antibody or hepatitis B surface antigen must have a negative polymerase chain reaction (PCR) result before enrollment; those who are PCR positive will be excluded
* Any uncontrolled active systemic infection
* Major surgery within 4 weeks of first dose of study drug
* Any life threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk
* Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to randomization
* Unable to swallow capsules or malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction
* Concomitant use of warfarin or other vitamin K antagonists
* Requires treatment with a strong cytochrome P450 (CYP) 3A4/5 inhibitor
* Lactating or pregnant
* Unwilling or unable to participate in all required study evaluations and procedures
* Unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local subject privacy regulations)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2021-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Coutre, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - City of Hope, Duarte, California
  - Stanford University, School of Medicine, Stanford, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Ibrutinib, Venetoclax)
Started | 22
Completed | 20
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ibrutinib, Venetoclax)
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (9.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 19
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR)
Description: Complete Response (CR) will be assessed as the number of participants who, based on investigator assessment based on the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria, achieve a complete remission. IWCLL complete remission is defined as follows.
  * Lymphadenopathy: none > 1.5 cm
  * Blood lymphocytes: < 4,000/µL
  * Hepatomegaly: none
  * Splenomegaly: none
  * Bone marrow: normocellular with < 30 lymphocytes, no B lymphoid nodules.
  The outcome is reported as the number of participants who achieve CR, a number without dispersion.
Time Frame: 62 weeks
Population: Some participants withdrew consent before the assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ibrutinib, Venetoclax)
Number analyzed (Participants) | 20
Participants | 12

2. Secondary Outcome: Duration of Response (DoR)
Description: Duration of response (DoR) refers to a participant maintaining clinical response after achieving either complete response (CR) or partial response (PR). The outcome is reported as the number of subjects who have maintained clinical response through 117 weeks. Response defined as the following.
  CR.
  * Lymphadenopathy: none > 1.5 cm
  * Blood lymphocytes: < 4,000/µL
  * Hepatomegaly: none
  * Splenomegaly: none
  * Bone marrow: normocellular with < 30 lymphocytes, no B lymphoid nodules. PR.
  * Lymphadenopathy: decrease ≥ 50%
  * Blood lymphocytes: decrease ≥ 50%
  * Hepatomegaly: decrease ≥ 50%
  * Splenomegaly: decrease ≥ 50%
  * Bone marrow: not considered.
Time Frame: 117 weeks
Population: Some participants withdrew consent before the assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ibrutinib, Venetoclax)
Number analyzed (Participants) | 17
Participants | 15

3. Secondary Outcome: Minimal Residual Disease (MRD)
Description: Minimal residual disease (MRD) refers to the small numbers of leukemic cells that can remain in the participant after treatment, and may not be associated with any symptoms (remission). Although the participant may feel "healthy," the MRD is a major cause of eventual leukemic relapse. "MRD-negative" is the ideal treatment outcome. MRD negativity was defined as less than one leukemic cell per 10,000 leukocytes as assessed by bone marrow-based flow cytometry. The outcome is reported as the number of participants who were positive for MRD, or negative.
Time Frame: 117 weeks
Population: Test results were not available for all participants. "Negligible" was considered as negative.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ibrutinib, Venetoclax)
Number analyzed (Participants) | 16
Participants
  Minimal residual disease (MRD)-negative | 13
  Minimal residual disease (MRD)-positive | 3

4. Secondary Outcome: Overall Response (OR)
Description: Overall response (OR) is the overall number of subjects that begin treatment and achieve a complete response (CR); partial response (PR); or Stable Disease (SD) 62 weeks after the beginning of treatment, according to the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria. IWCLL CR is defined as follows. The outcome is reported as the number of participants who achieve CR, PR, or SD, and number without dispersion.
  CR:
  * Lymphadenopathy: none > 1.5 cm
  * Blood lymphocytes: < 4,000/µL
  * Hepatomegaly: none
  * Splenomegaly: none
  * Bone marrow: normocellular with < 30 lymphocytes, no B lymphoid nodules.
  PR:
  * Lymphadenopathy: decrease ≥ 50%
  * Blood lymphocytes: decrease ≥ 50%
  * Hepatomegaly: decrease ≥ 50%
  * Splenomegaly: decrease ≥ 50%
  * Bone marrow: not considered.
  SD:
  * Lymphadenopathy: change of ± 49%
  * Blood lymphocytes: change of ± 49%
  * Hepatomegaly: change of ± 49%
  * Splenomegaly: change of ± 49%
  * Bone marrow: not considered.
Time Frame: 62 weeks
Population: Some participants withdrew before the assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ibrutinib, Venetoclax)
Number analyzed (Participants) | 20
Participants
  Complete Response (CR) | 12
  Partial Response (PR) | 8
  Stable Disease (SD) | 0

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) represents the amount of time the participants remain alive after treatment. The outcome is reported as the number of participants remaining alive at 117 weeks (about 2 years and 3 months) after the start of treatment, a number without dispersion.
Time Frame: Through 117 weeks
Population: Those participants who withdrew consent or were withdrawn for other medical treatments before 117 weeks are not included.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ibrutinib, Venetoclax)
Number analyzed (Participants) | 16
Participants | 16

6. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is a term that means to remain alive with progressive disease (PD). PD is defined as
  * Lymphadenopathy: Increase ≥ 50%
  * Blood lymphocytes: Increase ≥ 50%
  * Hepatomegaly: Increase ≥ 50%
  * Splenomegaly: Increase ≥ 50%
  * Bone marrow: not considered.
  The outcome is reported as the number of participants who remained alive without PD 117 weeks after the beginning of treatment.
Time Frame: 117 weeks
Population: Some participants withdrew consent before the assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ibrutinib, Venetoclax)
Number analyzed (Participants) | 17
Participants | 15

7. Secondary Outcome: Time-to-progression (TTP)
Description: Time-to-progression (TTP) is a measure of the length of time from the beginning of treatment until progressive disease (PD). PD is defined as
  * Lymphadenopathy: Increase ≥ 50%
  * Blood lymphocytes: Increase ≥ 50%
  * Hepatomegaly: Increase ≥ 50%
  * Splenomegaly: Increase ≥ 50%
  * Bone marrow: not considered.
  The outcome will be reported as the median TTP as determined by Kaplan-Meier methodology, with 95% confidence interval (95% CI).
Time Frame: Through 117 weeks
Population: An insufficient number of participants have experienced disease progression to determine a median value for that time period. This is expressed statistically as "Median Not Reached."
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ibrutinib, Venetoclax)
Number analyzed (Participants) | 17
months | NA [NA to NA] — An insufficient number of participants have experienced disease progression to determine a median value for that time period. This is expressed statistically as "Median Not Reached."

8. Other Pre Specified Outcome: Time-to-next-treatment (TTNT)
Description: The time-to-next-treatment (TTNT) is a measure of the period of time from the beginning of treatment until the patient has to receive a different treatment for his/her disease. TTNT was assessed as the time period until the participants next anti-chronic lymphocytic leukemia (CLL) treatment.
  The outcome will be reported as the median TTNT as determined by Kaplan-Meier methodology, with 95% confidence interval (95% CI).
Time Frame: Through 117 weeks
Population: An insufficient number of participants have advanced to a next treatment to determine a median value for that time period. This is expressed statistically as "Median Not Reached."
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ibrutinib, Venetoclax)
Number analyzed (Participants) | 17
months | NA [NA to NA] — An insufficient number of participants have advanced to a next treatment to determine a median value for that time period. This is expressed statistically as "Median Not Reached."

ADVERSE EVENTS:
Time Frame: 117 weeks
Arm/Group | Treatment (Ibrutinib, Venetoclax)
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 10/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ibrutinib, Venetoclax) (N=22)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Mastoiditis (Ear and labyrinth disorders) | 1 (1)
Fracture Skull (Injury, poisoning and procedural complications) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sepsis (Infections and infestations) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) -Other Hodgkins Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) -Other Squamous cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1)
Acute heart failure (Cardiac disorders) | 1 (1)
Aortic valve disease; Critical Stenosis (Cardiac disorders) | 1 (1)
Injury, poisoning and procedural complications - Other, Prostatectomy Pros (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ibrutinib, Venetoclax) (N=22)
Neutrophil count decreased (Investigations) | 19 (47)
Anemia (Blood and lymphatic system disorders) | 18 (45)
Leukocytosis (Blood and lymphatic system disorders) | 13 (16)
Lymphocyte count decreased (Investigations) | 8 (8)
Investigations - Other, Absolute monocyte (Investigations) | 3 (6)
Investigations - Other, Phosphorous level elevated (Investigations) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Ear and labyrinth disorders-Others, Tympanomastoidectomy (Ear and labyrinth disorders) | 1 (1)
Eye disorders-Other, Bilateral optic neuropathy (Eye disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Eye disorders-Other, cataracts, bilateral surgery (Eye disorders) | 3 (3)
Blurred vision (Eye disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 17 (26)
Nausea (Gastrointestinal disorders) | 11 (14)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7 (8)
Constipation (Gastrointestinal disorders) | 4 (4)
Mucositis oral (Gastrointestinal disorders) | 4 (4)
Gastrointestinal disorders-others, upper gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders-others, Oral stomatitis (Gastrointestinal disorders) | 1 (1)
Fatigue (Gastrointestinal disorders) | 10 (12)
Fever (Gastrointestinal disorders) | 3 (3)
Upper respiratory infection (Infections and infestations) | 9 (11)
Sinusitis (Infections and infestations) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Infections and Infestations, other, HSV (Infections and infestations) | 1 (1)
White blood cell decreased (Investigations) | 20 (41)
Platelet count decreased (Investigations) | 18 (33)
Creatinine increased (Investigations) | 6 (7)
Investigations. Other Lactate dehydrogenase increase (Investigations) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 10 (18)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (18)
Hyperphosphatemia (Metabolism and nutrition disorders) | 9 (9)
Blood bilirubin increased (Investigations) | 3 (5)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Metabolism and Nutrition disorders-Others. Hypogammaglobulinemia (Metabolism and nutrition disorders) | 5 (9)
Edema limbs (General disorders) | 8 (8)
Arthalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Peripheral Neuropathy (Nervous system disorders) | 1 (1)
Musculoskeletal and Connective Tissue Disorders, Other, Varicose veins (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps)-Others prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1)
Acute kidney Injury (Renal and urinary disorders) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 5 (8)
Chest pain (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Cardiac disorders-Other, ablation (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 13 (13)
Pruritis (Skin and subcutaneous tissue disorders) | 5 (6)
Rash (Skin and subcutaneous tissue disorders) | 5 (6)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 4 (4)
Skin and Subcutaneous Tissue Disorders-Other, Cellulitis (Skin and subcutaneous tissue disorders) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps)-Others, Lentigo melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin and Subcutaneous Tissue Disorders-Other, subcutaneous tissue disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and Subcutaneous Tissue Disorders-Other, Rosacea (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and Subcutaneous Tissue Disorders-Other, Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Paronychia (Infections and infestations) | 1 (1)
Aortic valve disease; Critical Stenosis (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT03045328/Prot_SAP_001.pdf
  • Informed Consent Form (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/28/NCT03045328/ICF_000.pdf